CLINICAL TRIAL: NCT01356355
Title: Double Blind Exploratory Three Arm Randomized Trial to Evaluate the Safety and Efficacy of Herbal Preparation 'Herbmed Plus' in Ureteral Stent Discomfort
Brief Title: Study of Herbmed Plus in Ureteral Stent Discomfort
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr .S.B.PATANKAR (Other)
Responsible Party: Sponsor-Investigator, Dr .S.B.PATANKAR, Amai Charitable Trust,ACE Hospital Pune, Amai Charitable Trust
Organization: Amai Charitable Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACE/HMP-02
Record Dates: First submitted 2011-05-16; First posted 2011-05-19 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Ureteral Stent Discomfort
Keywords: Stent discomfort; Herbmed plus; Tolterodine
MeSH Terms: interventions — Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Herbmed plus (Experimental): One capsule twice a day daily till ureteral stent in situ
  Interventions: Drug: Herbmed plus
- Placebo (Placebo Comparator): One capsule twice a day daily till ureteral stent in situ
  Interventions: Drug: Placebo
- Tolterodine (Active Comparator): One capsule twice a day daily till ureteral stent in situ
  Interventions: Drug: Tolterodine

INTERVENTIONS:
Drug: Herbmed plus — one capsule of herbmed plus orally twice a day with meals till the ureteral stent is in situ.
  Arms: Herbmed plus
Drug: Placebo — One capsule twice a day daily till ureteral stent in situ
  Other Names: sugar pills manufactured to mimic Herbmed plus
  Arms: Placebo
Drug: Tolterodine — One capsule twice a day daily till ureteral stent in situ
  Other Names: Torq SR; Terol LA
  Arms: Tolterodine

SUMMARY:
The purpose of this study is to compare the efficacy and safety of the Ayurvedic formulation ,Herbmed Plus against placebo and anti-cholinergic drugs in relieving the ureteral stent discomfort.

DETAILED DESCRIPTION:
* To evaluate the tolerability of ayurvedic preparation, Herbmed Plus in management of ureteral stent discomfort
* To know whether the ayurvedic preparation Herbmed Plus ,can reduce the requirement of analgesics or not
* To know whether the ayurvedic preparation ,Herbmed Plus can replace the use of analgesics/ anti cholinergics in relieving ureteral stent discomfort ?

ELIGIBILITY:
Inclusion Criteria:The following patients would be enrolled in the study:

1. Age 18-75 years (Both inclusive)
2. Absence of urinary tract infection
3. Absence of lower urinary tract symptoms
4. Absence of urethral catheter
5. Patients with unilateral/bilateral ureteral stentSize of the stent ranging from 4/16 to 6/26.
6. Patients of reproductive potential (males and females) and willing to use a reliable means of contraception (e.g. hormonal contraceptive patch, intrauterine device and physical barrier) throughout study participation.

7Able and willing to give written informed consent and comply with the requirements of the study protocol

Exclusion Criteria:

1. Patients having evidence of urinary tract infection.
2. Chronic medication with α-blockers or anticholinergics and severe complications during the procedure
3. Uncontrolled diabetes, hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction.
4. Any other urogenital disorders.
5. Liver dysfunction, defined as total bilirubin >1.5 x the upper limit of Normal (ULN),Aspartate aminotransferase (AST/SGOT) > 2.5 x ULN, or alanine aminotransferase (ALT/SGPT) >2.5 x ULN.
6. Kidney disease, including serum creatinine level >1.5 x ULN.
7. Subjects on herbal supplements (plant extracts preparations or herbal medicines etc.) within previous 3 months.
8. Participated in another clinical drug trial within 3 months before recruitment.
9. Pregnancy or breast feeding.
10. Evidence of significant uncontrolled concomitant disease which in the Investigator's opinion would preclude patient participation.
11. Currently active alcohol or drug abuse or history of alcohol or drug abuse within 24 weeks prior to baseline.
12. Patients with psychiatric illness or other condition that would limit compliance with study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-04; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Comparative study for Safety , Efficacy of Herbmed plus and tolterodine in management of ureteral stent discomfort. | 3weeks to 3 months
  -To compare the efficacy and safety of the Herbmed plus against placebo and anti-cholinergic drugs in relieving the ureteral stent discomfort viz.Dysuria, Urgency Frequency,Haematuria,Loin and suprapubic pain ,consumption of analgesics.

SECONDARY OUTCOMES:
Tolerability of herbmed plus in management of ureteral stent discomfort | 3 weeks to 3 months
  * To evaluate the tolerability of Herbmed Plus in management of ureteral stent discomfort
  * To know whether the Herbmed Plus can reduce the requirement of analgesics or not
  * To know whether the Herbmed Plus can replace the use of analgesics/ anti cholinergics in relieving ureteral stent discomfort ?

CONTACTS AND LOCATIONS:
Overall Officials: SURESH B PATANKAR, MS,MCH, Principal Investigator — AMAI CHARITABLE TRUST (AMAI CHARITABLE TRUST'S ACE HOSPITAL PUNE)
Locations (1):
- AMAI Charitable Trust's ACE Hospital Pune, Pune, Maharashtra, India

REFERENCES:
- [Background] Patankar S, Dobhada S, Bhansali M, Khaladkar S, Modi J. A prospective, randomized, controlled study to evaluate the efficacy and tolerability of Ayurvedic formulation "varuna and banana stem" in the management of urinary stones. J Altern Complement Med. 2008 Dec;14(10):1287-90. doi: 10.1089/acm.2008.0189. PMID 19040391